CLINICAL TRIAL: NCT04540419
Title: Multicenter, Randomized, Double Blind, Placebo Controlled Parallel Group Study Evaluating Efficacy, Reactogenicity and Safety of Recombinant Vaccine Ad5-nCoV Against Novel Coronavirus Infection in Adult Volunteers
Brief Title: Clinical Trial of Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) Against COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NPO Petrovax (Industry)
Collaborators: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Prometheus_Rus
Record Dates: First submitted 2020-08-17; First posted 2020-09-07 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ad5-nCoV single dose (Experimental): 375 subjects, Ad5-nCoV containing 5E10 vp, single dose
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- Placebo single dose (Placebo Comparator): 125 subjects, Placebo containing 0 vp, single dose
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) — Intramuscular administration
  Arms: Ad5-nCoV single dose
Biological: Placebo — Intramuscular administration
  Arms: Placebo single dose

SUMMARY:
This study is a phase III clinical trial to evaluate efficacy, reactogenicity and safety of the vaccine Ad5-nCoV compared with placebo in volunteers at the age from 18 to 85 years，with the randomized, double-blind design

DETAILED DESCRIPTION:
A total of 500 healthy adult volunteers at the age from 18 to 85 years will be randomized into two treatment (vaccination) groups in ratio 3:1 by double-blind design.

Volunteers in group 1 (n=375) will be administered a single dose of the vaccine Ad5-nCoV (5E10vp).

Volunteers in group 2 (n=125): will be administered a single dose of placebo. Vaccine Ad5-nCoV or placebo will be administered intramuscularly into the deltoid muscle of the arm at a single dose of 0.5 mL (1 prefilled syringe).

ELIGIBILITY:
Inclusion Criteria:

1. Presence of signed and dated Informed Consent of volunteer for participation in this study.
2. Men and women at the age of 18-85 years.
3. Bodyweight index 18.5-30.0 kg/m2.
4. The negative result of the test, performed by using PCR, for the presence of SARS-CoV-2 RNA at the stage of screening.
5. Negative result for anti-SARS-CoV-2 IgM and IgG antibodies at the stage of screening.
6. No history of the diagnosis COVID-19.
7. Absence of close contacts with individuals, suspicious for infection SARS-CoV-2, or individuals, in whom the diagnosis COVID-19 was confirmed in laboratory within the last 14 days.
8. Absence of signs of respiratory infection within the last 14 days.
9. Negative results of human immunodeficiency virus (HIV), syphilis, hepatitis B and hepatitis C tests.
10. According to historical data and results of screening examination, a volunteer has no diseases and/or conditions, which in view of Investigator, may influence the safety of volunteer participation and evaluation of study results.
11. Volunteer consent for using safe contraceptive methods through all the study.

Exclusion Criteria:

1. Positive history of allergy, drug intolerance, including increased sensibility to any of components of the test drug product, as well as the history of serious adverse events in the administration of vaccines (such as allergic reactions, respiratory disturbance, angioedema, stomach pain).
2. Axillary body temperature ≥37.1 °C at the time of screening/randomization.
3. Systolic blood pressure more than 139 mm Hg or less than 100 mm Hg and/or diastolic blood pressure more than 90 mm Hg or less than 60 mm Hg.
4. Clinical significant abnormal laboratory and/or instrumental parameters at screening examination.
5. Acute infectious diseases less than 4 weeks ahead of conduction of screening procedures.
6. Acute and acute course of chronic diseases of GIT, liver, kidneys, cardiovascular, respiratory, nervous and endocrine systems.
7. History of blood and hematopoietic organ diseases.
8. History of diabetes mellitus.
9. History of epilepsy, epileptic syndrome, seizures.
10. History of congenital and acquired immunodeficiency, HIV-infection, lymphoma, leukaemia, systemic lupus erythematosus, juvenile rheumatoid arthritis or other autoimmune diseases.
11. History malignancies.
12. Using immunotropic preparations (immunomodulators, immunostimulators, immunodepressants), antiallergic, cytotoxic preparations for more than 10 sequential days within the last 3 months (except for inhalant and local using glucocorticoids [GCS] or using specified preparations less than 4 weeks ahead of the screening.
13. Using immunoglobulin preparations or blood transfusion less than 3 months ahead of the screening.
14. Using antipyretics (including non-steroidal anti-inflammatory agents and anilides) within 24 hours ahead of randomization.
15. Blood donation or loss (≥450 mL of blood or plasma) less than 3 months ahead of the screening.
16. Vaccination within 6 mon. ahead of screening or reluctance to refuse from the administration of any other vaccine during the study.
17. Anamnestic data/data on alcoholism, narcomania, drug abuse, mental illnesses.
18. Major surgery planned within the nearest 6 months or underwent within the last 6 months ahead of the screening.
19. Carrying out of body piercing procedures, an appendix of tattoo less than 1 month ahead of conduction of screening procedures and through all the study.
20. Pregnancy or breast-feeding period.
21. Participation in another clinical study within 3 months ahead of the screening.
22. Psychic, physical and other reasons, not allowing a volunteer to adhere to conditions and procedures of Study Protocol.
23. Volunteers, who are Clinical Site staff.
24. Other reasons, not allowing the volunteer to take part in this study in view of the study physician.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Superiority of the vaccine Ad5-nCoV to placebo by the level of seroconversion | Day 28 after vaccination
  Proportion of subjects with four-fold and higher increment of anti-receptor-binding domain antibodies [receptor-binding domain, RBD] of S-protein SARS-CoV-2).

SECONDARY OUTCOMES:
Immunogenicity of the vaccine Ad5-nCoV compared with placebo (titer of SARS-CoV-2 antibodies) | Day 14, 28 and after 6 months after vaccination.
  Geometric mean titer of RBD и S-protein SARS-CoV-2 antibodies.
Immunogenicity of the vaccine Ad5-nCoV compared with placebo (level of seroconversion) | Day 14, 28 and after 6 months after vaccination.
  Level of seroconversion (proportion of persons with four-fold and higher increment of RBD и S-protein SARS-CoV-2 antibodies).
Immunogenicity of the vaccine Ad5-nCoV compared with placebo (rise of SARS-CoV-2 antibodies) | Day 14, 28 and after 6 months after vaccination.
  Geometric mean fold rise of RBD и S-protein SARS-CoV-2 antibodies.
Immunogenicity of the vaccine Ad5-nCoV compared with placebo (T-cell response) | Day 14, 28 and after 6 months after vaccination.
  Quantity of T-cells.
Frequency of confirmed COVID-19 | Within 6 months after vaccination (except for COVID-19 cases within 14 days after vaccination)
  Frequency of confirmed COVID-19 (confirmed case of COVID-19: presence of clinical signs and positive result of laboratory test for RNA of virus SARS-CoV-2) (exploratory analysis).
Frequency of confirmed cases of COVID-19, requiring hospitalization | Within 6 months after vaccination (except for COVID-19 cases within 14 days after vaccination)
  Frequency of confirmed cases of COVID-19, requiring hospitalization. (confirmed case of COVID-19: presence of clinical signs and positive result of laboratory test for RNA of virus SARS-CoV-2) (exploratory analysis).
Frequency of cases with severe course of COVID-19 | Within 6 months after vaccination (except for COVID-19 cases within 14 days after vaccination)
  Frequency of cases with severe course of COVID-19 (confirmed case of COVID-19: presence of clinical signs and positive result of laboratory test for RNA of virus SARS-CoV-2) (exploratory analysis).
Frequency of death due to COVID-19. | Within 6 months after vaccination (except for COVID-19 cases within 14 days after vaccination)
  Frequency of death due to COVID-19 (exploratory analysis).
Reactogenicity of the vaccine Ad5-nCoV compared with placebo | Day 0 (day of vaccination), Day 2, Day 7
  Frequency and character of general and local postvaccinal reactions.
Frequency and character of adverse events and serious adverse events. | Day 0 - Month 6
  Frequency and character of adverse events and serious adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on vital parameters (blood pressure) | Day -7-1 (Screening), Day 0, Day 2, Day 7, Day 14, Day 28, Month 6
  Results of evaluation of vital parameters:
  * Systolic blood pressure
  * Diastolic blood pressure The researcher evaluates each of the vital parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on vital parameters (heart rate) | Day -7-1 (Screening), Day 0, Day 2, Day 7, Day 14, Day 28, Month 6
  Results of evaluation of vital parameters:
  • Heart rate. The researcher evaluates each of the vital parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on vital parameters (respiratory rate) | Day -7-1 (Screening), Day 0, Day 2, Day 7, Day 14, Day 28, Month 6
  Results of evaluation of vital parameters:
  • Respiratory rate. The researcher evaluates each of the vital parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of physical examination | Day -7-1 (Screening), Day 0, Day 2, Day 7, Day 14, Day 28, Month 6
  Results of physical examination includes examination of organs and systems:
  General state Ears, nose, throat Skin and examination of the injection site The lymph nodes The cardiovascular system Respiratory system Nervous system Abdominal organs Kidneys and urinary system Musculoskeletal system.
  During the physical examination, the researcher evaluates each of the systems in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of electrocardiography (Heart rate) | Day -7-1 (Screening), Day 2
  Results of electrocardiography:
  • Heart rate (HR) The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of electrocardiography | Day -7-1 (Screening), Day 2
  Results of electrocardiography:
  * Intervals RR, PQ, QT
  * QRS complex
  * Corrected QT interval (QTcF). The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of serum chemistry (enzymes) | Day -7-1 (Screening), Day 2, Day 28
  Results of serum chemistry:
  alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), lactate dehydrogenase (LDH).
  The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of serum chemistry | Day -7-1 (Screening), Day 2, Day 28
  Results of serum chemistry:
  total bilirubin, creatinine, urea, fasting glucose. The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of serum chemistry | Day -7-1 (Screening), Day 2, Day 28
  Results of serum chemistry:
  total protein, C-reactive protein. The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of complete blood count (hemoglobin) | Day -7-1 (Screening), Day 2, Day 28
  Results of complete blood count: hemoglobin The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of complete blood count (hematocrit) | Day -7-1 (Screening), Day 2, Day 28
  Results of complete blood count: hematocrit.
  The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of complete blood count (erythrocytes) | Day -7-1 (Screening), Day 2, Day 28
  Results of complete blood count: erythrocytes.
  The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of complete blood count | Day -7-1 (Screening), Day 2, Day 28
  Results of complete blood count: platelets, leukocytes and leukocyte formula (neutrophils, lymphocytes, monocytes, eosinophils, basophils (absolute number).
  The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of complete blood count (erythrocyte sedimentation rate) | Day -7-1 (Screening), Day 2, Day 28
  Results of complete blood count: erythrocyte sedimentation rate
  The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of coagulogram | Day -7-1 (Screening), Day 2, Day 28
  Results of coagulogram:
  activated partial thromboplastin time, prothrombin time.
  The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of coagulogram (fibrinogen) | Day -7-1 (Screening), Day 2, Day 28
  Results of coagulogram: fibrinogen.
  The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of clinical urinalysis (relative density) | Day -7-1 (Screening), Day 2, Day 28
  Results of clinical urinalysis: relative density. The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of clinical urinalysis (pH) | Day -7-1 (Screening), Day 2, Day 28
  Results of clinical urinalysis: pH. The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of clinical urinalysis | Day -7-1 (Screening), Day 2, Day 28
  Results of clinical urinalysis: leukocytes, erythrocytes, cylinders . The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of clinical urinalysis (protein) | Day -7-1 (Screening), Day 2, Day 28
  Results of clinical urinalysis: protein . The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of clinical urinalysis (glucose) | Day -7-1 (Screening), Day 2, Day 28
  Results of clinical urinalysis:glucose . The researcher evaluates each of the parameter in the normal / abnormal categories. Clinically significant abnormalities should be reported as adverse events.
To evaluate safety of the vaccine Ad5-nCoV by its effect on results of determination of immunoglobulin E serum concentrations. | Day -7-1 (Screening), Day 28
  Results of determination of immunoglobulin E serum concentrations.

CONTACTS AND LOCATIONS:
Locations (7):
- Russia (7):
  - Federal budgetary institution of science "Central Research Institute of Epidemiology" of the Federal Service for Surveillance on Consumer Rights Protectionand Human Welfare, Moscow
  - State Budgetary Institution of Healthcare of the City of Moscow "City Polyclinic No. 2of the Department of Healthcare of the City of Moscow", Moscow
  - Federal State Autonomous Educational Institution of Higher Education "First MoscowState Medical University named after I.M. Sechenov "of the Ministry of Health of the Russian Federation, Moscow
  - Limited Liability Company "Research Center Eco-safety", Saint Petersburg
  - Federal State Budgetary Institution "Research Institute of Influenza named after A.A.Smorodintsev "of the Ministry of Health of the Russian Federation, Saint Petersburg
  - Private health care institution "Clinical hospital 'Russian Railways - Medicine' of the city of Yaroslavl", Yaroslavl
  - Municipal budgetary institution "Central City Hospital No. 7", Yekaterinburg

REFERENCES:
- [Derived] Lioznov D, Amosova I, Sheetikov SA, Zornikova KV, Serdyuk Y, Efimov GA, Tsyferov M, Khmelevskii M, Afanasiev A, Khomyakova N, Zubkov D, Tikhonov A, Zhu T, Barreto L, Dzutseva V. Immunogenicity and safety of a recombinant adenovirus type-5 COVID-19 vaccine in adults: Data from a randomised, double-blind, placebo-controlled, single-dose, phase 3 trial in Russia. PLoS One. 2023 Mar 8;18(3):e0278878. doi: 10.1371/journal.pone.0278878. eCollection 2023. PMID 36888640